CLINICAL TRIAL: NCT00670982
Title: Phase 2 Study of Bevacizumab in Combination With Vinorelbine and Trastuzumab for HER2-Positive, Metastatic Breast Cancer
Brief Title: Bevacizumab in Combination With Vinorelbine and Trastuzumab for HER2-Positive, Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Harold J. Burstein, MD, PhD (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); Genentech, Inc. (Industry); New Hampshire Oncology-Hematology PA (Unknown); Lowell General Hospital (Other); Hartford Hospital (Other)
Responsible Party: Sponsor-Investigator, Harold J. Burstein, MD, PhD, Associate Professor of Medicine, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-214
Record Dates: First submitted 2008-04-29; First posted 2008-05-02 (Estimated); Results first posted 2013-05-13 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer
Keywords: HER2 positive; bevacizumab; vinorelbine; trastuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Vinorelbine; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- First line treatment (Experimental): Patients with no prior therapy for metastatic breast cancer will receive bevacizumab intravenously every 2 weeks and vinorelbine intravenously once per week, and trastuzumab intravenously once per week
  Interventions: Drug: bevacizumab; Drug: vinorelbine; Drug: trastuzumab
- Second line treatment (Experimental): Patients with 1 prior line for metastatic breast cancer will receive bevacizumab intravenously every two weeks, vinorelbine intravenously once per week, and trastuzumab intravenously once per week.
  Interventions: Drug: bevacizumab; Drug: vinorelbine; Drug: trastuzumab

INTERVENTIONS:
Drug: bevacizumab — Given intravenously every 2 weeks
  Other Names: Avastin
Drug: vinorelbine — Given intravenously once a week
  Other Names: Navelbine
Drug: trastuzumab — Given intravenously once a week
  Other Names: Herceptin

SUMMARY:
The purpose of this research study is to determine the effects of the combination of bevacizumab, vinorelbine, and trastuzumab on participants and their cancer.

DETAILED DESCRIPTION:
* Participants will receive bevacizumab intravenously every 2 weeks. They will also receive trastuzumab and vinorelbine intravenously once a week. Therefore, treatments will alternate between receiving all three drugs (1st week, third week, fifth week, etc.) and receiving only trastuzumab and vinorelbine (2nd week, fourth week, sixth week, etc.) A treatment cycle lasts four weeks.
* During all treatment cycles a physical exam will be performed and the participant will be asked general health and specific questions about any problems they are experiencing.
* X-ray, CT scans, and/or MRI scans will be performed every 8 weeks (every 2 cycles) in order to assess the effect of the study treatment on the participants cancer. These tests are considered standard of care in patients receiving chemotherapy.
* Once a week blood counts will be performed and at least every 4 weeks, chemistry and other tests to measure any additional effect of the study drug and disease status will be checked. These tests are also considered standard of care for patients receiving chemotherapy.
* At the beginning of the study and at the 4- and 8-week time point, additional blood will be drawn in order to conduct research blood tests to measure the presence of cancer cells in the blood.
* A urine test and MUGA scan or echocardiogram will be done every 8 weeks while the participant in on the study.
* Participants can remain on the research study as long as the study treatment appears to be working and they are not experiencing unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive breast cancer, with metastatic disease.
* HER2-positive tumor
* Measurable disease defined as at least one lesion that can be accurately measured in at least one dimension as 20mm or greater with conventional techniques or as 10mm or greater with spiral CT scan
* 18 years of age or older
* Life expectancy of more than 12 weeks
* ECOG Performance Status of 0 or 1
* Normal organ and marrow function as outlined in the protocol
* Left ventricular ejection fraction 50% or greater as determined by RVG or echocardiogram within 30 days prior to initiation of protocol therapy
* Patients with stable or previously treated CNS metastases are eligible for study participation, provided there is no history of clinically significant CNS bleeding
* Men and women of child-bearing potential must agree to use adequate contraception prior to study entry and for the duration of study participation

COHORT A:

* No prior chemotherapy for treatment of metastatic breast cancer
* May NOT have received prior treatment with trastuzumab for recurrent or metastatic breast cancer
* No prior vinorelbine for treatment of breast cancer
* No prior bevacizumab for treatment of breast cancer
* May have received prior radiation therapy and/or any number of lines of hormonal therapy
* Prior trastuzumab therapy in the adjuvant setting is also allowed, providing that relapse occured at least 12 months following the last dose
* Must have recovered from all reversible toxicities related to prior therapy and may not have any pre-existing treatment-related toxicities in excess of Grade 1. Patients must have stopped prior radiation therapy at least 7 days prior to beginning protocol treatment

COHORT B:

* One prior line of chemotherapy for treatment of metastatic breast cancer or recurrence of breast cancer within 12 months of completion of adjuvant trastuzumab
* No prior vinorelbine for treatment of breast cancer
* No prior bevacizumab for treatment of breast cancer
* May have received prior radiation therapy and/or any number of lines of hormonal therapy
* Must have recovered from all reversible toxicities related to prior therapy and may not have any pre-existing treatment-related toxicities in excess of Grade 1. Patients must have stopped prior radiation therapy at least 7 days prior to beginning protocol treatment

Exclusion Criteria:

* Patients who have had chemotherapy within 14 days prior to entering the study, ot those who have not recovered adequately from adverse events due to agents administered earlier
* Concurrent radiation therapy
* History of Grade 3 or 4 allergic reactions attributed to compounds of similar chemical or biologic composition as the agents used in this study
* Prior therapy with bevacizumab or vinorelbine
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study
* Inadequately controlled hypertension
* Prior history of hypertensive crisis of hypertensive encephalopathy
* NHYA Grade II or greater congestive heart failure
* History of myocardial infarction of unstable angina within 6 months prior to study enrollment
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Progressive or untreated CNS metastases
* Significant vascular disease within 6 months prior to study enrollment
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of vascular access device, within 7 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria at screening
* Pregnant or lactating
* Current and ongoing treatment with full-dose warfarin or its equivalent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-05; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold J. Burstein, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (7):
- United States (7):
  - Hartford Hospital, Hartford, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Faulkner Hospital, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - New Hampshire Oncology-Hematology PA, Hooksett, New Hampshire

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between May 2008 and March 2010.
Groups:
- First Line Treatment: Patients with no prior therapy for metastatic breast cancer will receive bevacizumab(10mg/kg) intravenously every 2 weeks and vinorelbine(25mg/m2) intravenously once per week, and trastuzumab (4 mg/kg) intravenously once per week
- Second Line Treatment: Patients with 1 prior line for metastatic breast cancer will receive bevacizumab(10mg/kg) intravenously every two weeks, vinorelbine (25mg/m2) intravenously once per week, and trastuzumab(4 mg/kg) intravenously once per week.
Period: Overall Study
Arm/Group | First Line Treatment | Second Line Treatment
Started | 22 | 7
Completed | 22 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | First Line Treatment | Second Line Treatment | Total
Number analyzed (Participants) | 22 | 7 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 7 | 29
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 51.5 (8) | 46.7 (6.9) | 50.3 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 7 | 29
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 7 | 29

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Alive and Without Progression of Disease at 1 Year From Start of Protocol-based Therapy.
Description: Percentage of patients on study without progression at one year after first treatment on study.The date of progression was defined as the earliest occurence of any of the following events: progressive disease by RECIST v1.0, date of initiation of new anticancer therapy, or death due to any cause. New anticancer therapy was defined as the addition or initiation of any new agent for treatment of cancer not including trastuzumab, vinorelbine or bevacizumab.
Time Frame: 1 year
Population: What percentage of patients were still on study and without progression at one year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | First Line Treatment | Second Line Treatment
Number analyzed (Participants) | 22 | 7
percentage of participants | 36 [17 to 59] | 29 [4 to 71]

2. Secondary Outcome: Objective Response Rate
Description: Objective response rate by Response Evaluation Criteria in Solid Tumors (RECIST v1.0) and assessed by computed tomography.Complete response (CR), disappearance of all target and non-target lesions; partial response (PR), >/=30% decrease in the sum of longest dimensions of target lesions; objective response rate = CR + PR.
Time Frame: 1 year
Population: Confirmed objective response rate
Measure: Number; unit: percentage of participants
Arm/Group | First Line Treatment | Second Line Treatment
Number analyzed (Participants) | 22 | 7
percentage of participants | 73 | 71

3. Secondary Outcome: Progression-free Survival
Description: Median progression free survival measured in months
Time Frame: 3 years
Population: Median time from registration to progression of disease
Measure: Median (Full Range); unit: months
Arm/Group | First Line Treatment | Second Line Treatment
Number analyzed (Participants) | 22 | 7
months | 9.9 [1.6 to 22.3] | 7.8 [3.5 to 22.0]

ADVERSE EVENTS:
Time Frame: 3 years
Description: Since all patients received the same study treatment, all adverse events were collected and reported together.
Groups:
- All Study Participants: All participants received the same study treatment, so cumulative adverse events are reported here.
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 9/29
Other Adverse Events (participants affected / at risk) | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=29)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Cerebrovascular Ischemia (Vascular disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 5 (9)
Perforated Appendix (Gastrointestinal disorders) | 1 (1)
Surgical Intervention (Surgical and medical procedures) | 1 (1)
Cataracts (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=29)
Abdominal Pain (Gastrointestinal disorders) | 5 (8)
Alkaline Phosphatase (Blood and lymphatic system disorders) | 6 (23)
Allergic Reaction (General disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (39)
ALT-SPGT or AST-SGOT (Hepatobiliary disorders) | 23 (130)
Anorexia (Gastrointestinal disorders) | 9 (20)
Bone-pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bleeding (Blood and lymphatic system disorders) | 6 (10)
Cataract (Eye disorders) | 5 (6)
Chest wall-pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Constipation (Gastrointestinal disorders) | 15 (48)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (14)
Dehydration (General disorders) | 3 (3)
Depression (Psychiatric disorders) | 2 (3)
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 14 (38)
Dizziness (Nervous system disorders) | 2 (4)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dyspnoea (Gastrointestinal disorders) | 5 (8)
Extremity-limb-pain (Musculoskeletal and connective tissue disorders) | 8 (14)
Fatigue (General disorders) | 27 (164)
Febrile Neutropenia (Blood and lymphatic system disorders) | 6 (8)
Fever without Neutropenia (General disorders) | 13 (26)
GI-other (Gastrointestinal disorders) | 2 (2)
Head/headache (Nervous system disorders) | 15 (25)
Hemoglobin (Blood and lymphatic system disorders) | 27 (226)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Endocrine disorders) | 14 (43)
Hypernatremia (Metabolism and nutrition disorders) | 2 (3)
Hypertension (Blood and lymphatic system disorders) | 11 (56)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (17)
Hypokalemia (Metabolism and nutrition disorders) | 4 (9)
Hyponatremia (Metabolism and nutrition disorders) | 6 (6)
Infection (Infections and infestations) | 7 (15)
Insomnia (General disorders) | 5 (8)
Joint-pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Leukocytes (Blood and lymphatic system disorders) | 24 (144)
Lymphopenia (Blood and lymphatic system disorders) | 3 (4)
Metabolic/Laboratory-other (Metabolism and nutrition disorders) | 4 (6)
Muco/stomatitis (Infections and infestations) | 10 (12)
Muscle-pain (Musculoskeletal and connective tissue disorders) | 6 (9)
Nasal cavity/paranasal sinus reaction (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 15 (52)
Neurologic-other (Nervous system disorders) | 3 (5)
Neuropathy-motor (Nervous system disorders) | 8 (8)
Neuropathy-sensory (Nervous system disorders) | 16 (71)
Neutrophils (Blood and lymphatic system disorders) | 28 (201)
Nose-hemorrhage (Blood and lymphatic system disorders) | 16 (49)
Ocular (Eye disorders) | 2 (3)
Oral cavity-hemorrhage (Blood and lymphatic system disorders) | 2 (3)
Pain-other (Nervous system disorders) | 2 (3)
Platelets (Blood and lymphatic system disorders) | 3 (4)
Proteinuria (Renal and urinary disorders) | 6 (24)
Pruitus/itching (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (4)
Rigors (General disorders) | 4 (5)
Taste disturbance (General disorders) | 2 (2)
Throat/pharynx/larynx-pain (Nervous system disorders) | 3 (4)
Tinnitus (Ear and labyrinth disorders) | 2 (3)
Voice changes /dysarthria (General disorders) | 5 (9)
Vomiting (Gastrointestinal disorders) | 10 (14)
weight-loss (General disorders) | 3 (5)
wound-non infectious (General disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No